CLINICAL TRIAL: NCT02534207
Title: A Single-Centre, Non-Randomised, Open Label, Positron Emission Tomography Imaging Study to Assess Occupancy of α5-Containing GABAA Receptors by RO5186582 in Healthy Volunteers of Japanese Origin
Brief Title: Basmisanil Positron Emission Tomography Study in Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BP29784; 2015-001621-16 (EudraCT Number)
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — basmisanil

ARMS (1):
- Basmisanil in Japanese Healthy Volunteers (Experimental): Japanese healthy volunteers will receive a single oral dose of RO5186582 within 15 minutes after completing a standard meal.
  Interventions: Drug: Basmisanil

INTERVENTIONS:
Drug: Basmisanil — Single oral dose: Basmisanil doses between 20 milligrams (mg) and 960 mg may be used in this study. The planned doses for the first two participants are 160 mg and 480 mg, respectively. Basmisanil dose for subsequent participants will be decided by the investigator and sponsor during the study, based on on-going review of emerging data.
  Other Names: RO5186582, RG1662

SUMMARY:
This study will evaluate the relationship between basmisanil plasma concentrations and the occupancy of Gamma-Amino Butyric Acid A (GABAA) receptor subtypes containing an alpha5 (α5) subunit in healthy Japanese volunteers. Each participant will have two post-screening imaging sessions. In the first imaging session, participants will have a baseline Positron Emission Tomography (PET) scan. In the second imaging session, participants will receive a single oral dose of basmisanil, followed by two on-treatment PET scans at about 4 and 10 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese healthy volunteer, who was born in Japan, has 4 ethnically Japanese grandparents and has lived outside Japan for no longer than 5 years
* A body mass index (BMI, Quetelet index) in the range 18.0 to 32.0 kilograms per square meter (kg/m^2)
* Willingness and ability to comply with study restrictions

Exclusion Criteria:

* A history of epilepsy, convulsions or significant head injury, or other structural brain abnormality
* Pregnant or lactating or not using acceptable contraception
* Presence or history of severe adverse reaction to any drug or a history of sensitivity to basmisanil or the PET radioligand (RO15-4513)
* Significant exposure to radiation within the previous 12 months
* Any other clinically relevant abnormalities, concomitant diseases or ongoing medical conditions

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Brain α5 Subunit-Containing GABAA Receptors Occupied by Basmisanil (Receptor Occupancy) Following a Single Dose of Basmisanil in Selected Regions of Interest (ROIs) Assessed by PET Imaging | Day 1
Correlation Between Basmisanil Plasma Concentration and Occupancy of Brain α5 Subunit-Containing GABAA Receptors | Day 1

SECONDARY OUTCOMES:
Brain GABAA Receptor α5 Subunit Levels in Selected ROIs Assessed by PET Imaging | Day 1
Percentage of Participants With Adverse Events | From Baseline up to 7-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United Kingdom (3):
  - Hammersmith Medicines Research; Central Middlesex Hospital, London
  - London
  - Imanova Limited, London